CLINICAL TRIAL: NCT06456346
Title: A Phase 3, Randomized, Double-blind, Active-Comparator-Controlled Clinical Study to Evaluate the Efficacy and Safety of Bomedemstat (MK-3543) Versus Hydroxyurea in Cytoreductive Therapy Naïve Essential Thrombocythemia Participants
Brief Title: Bomedemstat vs Hydroxyurea for Essential Thrombocythemia (MK-3543-007)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3543-007; 2023-505232-36-00 (Registry Identifier: EU CT); MK-3543-007 (Other: MSD); jRCT2031240181 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); U1111-1290-8287 (Registry Identifier: UTN)
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Essential Thrombocythemia
Keywords: essential thrombocythemia; ET; bomedemstat; IMG-7289
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — bomedemstat; Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bomedemstat (Experimental): Participants will receive active bomedemstat and hydroxyurea placebo daily for up to approximately 52 weeks. Dosage will be adjusted either up or down within specified time parameters for each participant to the dose that provides sufficient exposure to safely inhibit thrombopoiesis to decrease platelet counts to the target range. Participants who complete treatment at Week 52 will be eligible to continue treatment in the extended treatment phase. Unblinding will occur and placebo discontinued once all participants have completed at least 52 weeks of therapy or otherwise discontinued.
  Interventions: Drug: Bomedemstat; Drug: Hydroxyurea placebo
- Hydroxyurea (Active Comparator): Participants will receive active hydroxyurea and bomedemstat placebo daily for up to 52 weeks. Dosage will be adjusted either up or down within specified time parameters for each participant to the dose that provides sufficient exposure to safely inhibit thrombopoiesis to decrease platelet counts to the target range. Participants who complete treatment at Week 52 will be eligible to continue treatment in the extended treatment phase. Unblinding will occur and placebo discontinued once all participants have completed at least 52 weeks of therapy or otherwise discontinued.
  Interventions: Drug: Hydroxyurea; Drug: Bomedemstat placebo

INTERVENTIONS:
Drug: Bomedemstat — Oral capsule
  Other Names: MK-3543; IMG-7289
  Arms: Bomedemstat
Drug: Hydroxyurea — Oral capsule
  Arms: Hydroxyurea
Drug: Bomedemstat placebo — Oral capsule placebo
  Arms: Hydroxyurea
Drug: Hydroxyurea placebo — Oral capsule placebo
  Arms: Bomedemstat

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of bomedemstat compared with hydroxyurea in cytoreductive therapy naïve essential thrombocythemia (ET) participants for whom cytoreductive therapy is indicated. Its primary objective is to compare bomedemstat to hydroxyurea with respect to durable clinicohematologic response (DCHR). The primary hypothesis is that bomedemstat is superior to hydroxyurea with respect to DCHR.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Essential Thrombocythemia (ET) based on World Health Organization Criteria for myeloproliferative neoplasms, and an indication for cytoreductive therapy regardless of age or risk status
* Has a centrally assessed bone marrow fibrosis score of Grade 0 or Grade 1, as per a modified version of the European Consensus Criteria for Grading Myelofibrosis
* Has received no prior cytoreductive treatment for their ET
* Human Immunodeficiency Virus (HIV)-infected participants have well controlled HIV on antiretroviral therapy
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load
* Participants with history of Hepatitis C Virus (HCV) infection are eligible if HCV viral load is undetectable

Exclusion Criteria:

* History of any illness/impairment of gastrointestinal function that might interfere with drug absorption
* History of a malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has an active infection requiring systemic therapy
* Has had a major surgery <4 weeks prior to first dose of study intervention or has not recovered from side effects of major surgery >4 weeks prior to first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2027-09-28 (Estimated); Study Completion 2028-03-24 (Estimated)

PRIMARY OUTCOMES:
Durable Clinicohematologic Response (DCHR) Rate | Up to Week 52
  DCHR rate is the percentage of participants with DCHR, defined as a confirmed reduction of platelet count to ≤400 × 10^9/L, absence of white blood cell (WBC) count elevation to >10 × 10^9/L locally assessed to be due to ET, starting by Week 24 and maintained for at least 24 weeks, and the absence of any thrombotic or major hemorrhagic events or disease progression to myelofibrosis (MF), myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) by Week 52.

SECONDARY OUTCOMES:
Change From Baseline in Myelofibrosis Symptom Assessment Form version 4.0 (MFSAF v4.0) Individual Fatigue Symptom Item Score | Baseline and pre-specified timepoints up to Week 52
  The MFSAF v4.0 is a 7-item participant-reported myelofibrosis symptom assessment which asks respondents to report symptom severity at its worst for each of the 7 items on a 0 (Absent) to 10 (Worst Imaginable) numeric rating scale.
Change From Baseline in Patient-reported Outcomes Measurement Information System (PROMIS) Fatigue SF-7a Total Fatigue Score | Baseline and pre-specified timepoints up to Week 52
  The PROMIS F SF-7a is a 7-item participant-reported assessment that measures both the experience of fatigue and the interference of fatigue on daily activities over the past week. Response options are on a 5-point Likert scale, ranging from 1 = never to 5 = always.
Change From Baseline in MFSAF v4.0 Total Symptom Score | Baseline and Week 52
  The MFSAF v4.0 is a 7-item participant-reported myelofibrosis symptom assessment which asks respondents to report symptom severity at its worst for each of the 7 items on a 0 (Absent) to 10 (Worst Imaginable) numeric rating scale. The change from baseline in MFSAF total score for all symptoms will be presented.
Duration of Hematologic Remission (DOHR) | Up to Week 52
  For participants who demonstrate hematologic remission, DOHR is defined as the time from the first documented evidence of platelet and WBC counts reduction until platelet or WBC counts increase to above acceptable threshold.
Number of Participants Who Experience Thrombotic Events | Up to approximately 52 weeks
  Thrombotic events include but are not limited to new or recurrent acute myocardial infarction, unstable angina, stroke, transient ischemic attack, deep venous thrombosis, pulmonary embolism, thrombotic digital ischemia, or other thrombotic events.
Number of Participants Who Experience Major Hemorrhagic Events | Up to approximately 52 weeks
  Major hemorrhagic events include but are not limited to fatal bleeding, and/or symptomatic bleeding in a critical area or organ such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a decrease in hemoglobin level of 2 g/dL or more, or leading to transfusion of 2 or more units of whole blood or red cells.
Disease Progression Rate | Up to Week 52
  Disease progression rate is the percentage of participants with disease progression, defined as the transformation to post-essential thrombocythemia myelofibrosis, myelodysplastic syndrome, or AML as assessed by the adjudication committee.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (163):
- United States (15):
  - Palo Verde Cancer Specialists ( Site 0052), Glendale, Arizona
  - Los Angeles Cancer Network ( Site 0025), Glendale, California
  - Stanford Cancer Center ( Site 0024), Palo Alto, California
  - Exempla Lutheran Medical Center ( Site 0014), Golden, Colorado
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0006), Fort Wayne, Indiana
  - University of Michigan ( Site 0003), Ann Arbor, Michigan
  - Levine Cancer Institute ( Site 0009), Charlotte, North Carolina
  - Duke University Health System (DUHS) ( Site 0012), Durham, North Carolina
  - Wake Forest Baptist Health-Internal Medicine, Section on Hematology & Oncology ( Site 0013), Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center ( Site 0028), Columbus, Ohio
  - Oregon Health & Science University ( Site 0018), Portland, Oregon
  - University of Texas MD Anderson Cancer Center ( Site 0026), Houston, Texas
  - University of Texas Health Science Center at San Antonio ( Site 0021), San Antonio, Texas
  - University of Virginia ( Site 0020), Charlottesville, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 0008), Richmond, Virginia
- Argentina (4):
  - Hospital Universitario Austral ( Site 0101), Pilar, Buenos Aires
  - Hospital Italiano de Buenos Aires ( Site 0102), ABB, Buenos Aires F.D.
  - C.I.C.E. 9 de Julio ( Site 0104), San Miguel de Tucumán, Tucumán Province
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares ( Site 0105), Santa Fe
- Australia (5):
  - Westmead Hospital ( Site 0201), Westmead, New South Wales
  - Royal Adelaide Hospital-Haematology Clinical Trials Unit ( Site 0203), Adelaide, South Australia
  - Monash Health-Haematology Research ( Site 0202), Clayton, Victoria
  - Austin Health-Cancer Clinical Trials Centre ( Site 0206), Heidelberg, Victoria
  - Royal Perth Hospital-Haematology ( Site 0204), Perth, Western Australia
- Ordensklinikum Linz GmbH Elisabethinen ( Site 0562), Linz, Upper Austria, Austria
- Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre ( Site 0037), Greenfield Park, Quebec, Canada
- Chile (6):
  - IC La Serena Research ( Site 0150), La Serena, Coquimbo Region
  - FALP-UIDO ( Site 0148), Santiago, Region M. de Santiago
  - Clínica Inmunocel ( Site 0147), Santiago, Region M. de Santiago
  - Clínica Alemana de Santiago ( Site 0143), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0142), Santiago, Region M. de Santiago
  - Biocenter ( Site 0149), Concepción, Región del Biobío
- China (24):
  - The First Afflilated Hospital of Bengbu Medical College ( Site 0651), Bengbu, Anhui
  - Anhui Provincial Hospital ( Site 0657), Hefei, Anhui
  - Peking University Third Hospital-Hematology ( Site 0659), Beijing, Beijing Municipality
  - Chinese Academy of medical science, Peking Union Medical College Hospital(Dongdan) ( Site 0675), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 0666), Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Fujian Medical University ( Site 0671), Quanzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 0658), Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University-hematology department ( Site 0668), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital-Department of Hematopathology ( Site 0655), Guangzhou, Guangdong
  - The Second Afilliated Hospital of Hebei Medical University ( Site 0650), Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University ( Site 0649), Shijiazhuang, Hebei
  - Henan Cancer Hospital-hematology department ( Site 0644), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 0642), Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University ( Site 0676), Suzhou, Jiangsu
  - The First affiliated hospital of Nanchang University (Xianghu campus) ( Site 0645), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Hematology ( Site 0672), Changchun, Jilin
  - Shaanxi provincial people's hospital ( Site 0652), Xi'an, Shaanxi
  - Jinan Central Hospital ( Site 0667), Jinan, Shandong
  - Zhongshan Hospital,Fudan University-Hematology ( Site 0674), Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University ( Site 0669), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 0661), Chengdu, Sichuan
  - Institute of hematology&blood disease hospital-Hematology ( Site 0641), Tianjin, Tianjin Municipality
  - The first Affiliated Hospital, Zhejiang University School of Medicine ( Site 0646), Hangzhou, Zhejiang
  - Zhejiang University School of Medicine-The Fourth Affiliated Hospital ( Site 0662), Yiwu, Zhejiang
- Colombia (3):
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 0164), Medellín, Antioquia
  - Los Cobos Medical Center ( Site 0165), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 0162), Montería, Departamento de Córdoba
- Denmark (4):
  - Rigshospitalet-Hematology - CTU ( Site 0321), Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby-Blodsygdomme ( Site 0324), Aarhus, Central Jutland
  - Roskilde Sygehus-Department of Hematology ( Site 0323), Roskilde, Region Sjælland
  - Odense Universitetshospital-Department of Hematology ( Site 0325), Odense C, Region Syddanmark
- France (10):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet-Hematology ( Site 0349), Nice, Alpes-Maritimes
  - CHU Bordeaux Haut-Leveque-service de mèdecine interne et maladies infectieuses ( Site 0346), Pessac, Aquitaine
  - Hôpital de la Conception ( Site 0351), Marseille, Bouches-du-Rhone
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE ( Site 0352), Toulouse, Haute-Garonne
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren ( Site 0344), Limoges, Haute-Vienne
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital-Hématologie et Thérapie Cellulaire ( Site 0342), Tours, Indre-et-Loire
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu ( Site 0347), Nantes, Loire-Atlantique
  - centre hospitalier lyon sud ( Site 0343), Pierre-Bénite, Rhone
  - HENRI MONDOR HOSPITAL ( Site 0348), Créteil, Val-de-Marne
  - Hopital Saint-Louis ( Site 0341), Paris
- Germany (8):
  - VK&K Studien GbR ( Site 0370), Landshut, Bavaria
  - Medizinische Hochschule Hannover ( Site 0371), Hanover, Lower Saxony
  - Universitätsklinikum Aachen ( Site 0367), Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 0366), Essen, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz-3. Medizinische Klinik und Poliklinik ( Site 0365), Mainz, Rhineland-Palatinate
  - Universitätsklinikum Halle ( Site 0361), Halle, Saxony-Anhalt
  - Universitätsklinikum Jena-Klinik für Innere Medizin II, Abt. Hämatologie und Internistische Onkolog ( Site 0364), Jena, Thuringia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0369), Berlin
- Queen Mary Hospital ( Site 0221), Hksar, Hong Kong
- Hungary (5):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Belgyógyászati Klinika ( Site 0407), Szeged, Csongrád megye
  - Petz Aladar Egyetemi Oktato Korhaz-Hematológia ( Site 0405), Győr, Győr-Moson-Sopron
  - Somogy Vármegyei Kaposi Mór Oktató Kórház-Haematológiai osztály ( Site 0406), Kaposvár, Somogy County
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókór-Haematológia osztály ( Site 0404), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Debreceni Egyetem Klinikai Kozpont-Belgyógyászati Klinika (Haematologia) ( Site 0402), Debrecen
- Israel (9):
  - Soroka Medical Center ( Site 0427), Beersheba
  - Rambam Health Care Campus ( Site 0429), Haifa
  - Carmel Hospital ( Site 0426), Haifa
  - Hadassah Medical Center ( Site 0424), Jerusalem
  - Galilee Medical Center ( Site 0431), Nahariya
  - Rabin Medical Center ( Site 0425), Petah Tikva
  - Sheba Medical Center ( Site 0428), Ramat Gan
  - Sourasky Medical Center ( Site 0422), Tel Aviv
  - Yitzhak Shamir Medical Center. ( Site 0421), Ẕerifin
- Italy (7):
  - Azienda Ospedaliero-Universitaria SS. Antonio e Biagio e Cesare Arrigo ( Site 0443), Alessandria, Ancona
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico ( Site 0447), Milan, Lombardy
  - Azienda Ospedaliera Universitaria Careggi ( Site 0441), Florence, Tuscany
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 0446), Bologna
  - Fondazione IRCCS Policlinico San Matteo-Oncology ( Site 0444), Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 0445), Roma
  - Ospedale di Circolo e Fondazione Macchi Varese ( Site 0442), Varese
- Japan (16):
  - Fujita Health University Hospital ( Site 0613), Toyoake, Aichi-ken
  - Ehime University Hospital ( Site 0612), Tōon, Ehime
  - Hokkaido University Hospital ( Site 0601), Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital ( Site 0603), Kobe, Hyōgo
  - Kanazawa University Hospital ( Site 0614), Kanazawa, Ishikawa-ken
  - Mie University Hospital ( Site 0615), Tsu, Mie-ken
  - National Hospital Organization Sendai Medical Center ( Site 0617), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 0607), Hirakata, Osaka
  - Kindai University Hospital ( Site 0600), Sakai, Osaka
  - Juntendo University Hospital ( Site 0611), Bunkyo-ku, Tokyo
  - University of Yamanashi Hospital ( Site 0606), Chūō, Yamanashi
  - Kyushu University Hospital ( Site 0605), Fukuoka
  - Fukushima Medical University Hospital ( Site 0616), Fukushima
  - University of Miyazaki Hospital ( Site 0609), Miyazaki
  - Okayama University Hospital ( Site 0604), Okayama
  - Nippon Medical School Hospital ( Site 0608), Tokyo
- Mexico (3):
  - Medivest Centro de Investigación Integral ( Site 0183), Chihuahua City, Chihuahua
  - Higiea Oncologia ( Site 0184), Mexico City, Mexico City
  - Centro de Investigacion Clinica de Oaxaca ( Site 0181), Oaxaca City, Oaxaca
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie-Oddział Hematoonkologii, Transplantacji Szp ( Site 0463), Lublin, Lublin Voivodeship
  - Pratia Onkologia Katowice ( Site 0461), Katowice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Hematologii i Transplantacji S ( Site 0466), Kielce, Świętokrzyskie Voivodeship
- Spain (10):
  - Hospital Germans Trias i Pujol-Instituto Catalán de Oncología de Badalona ( Site 0490), Badalona, Barcelona
  - Hospital Universitario Marqués de Valdecilla-Haematology ( Site 0486), Santander, Cantabria
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 0481), Barcelona, Catalonia
  - Institut Català d'Oncologia - L'Hospitalet ( Site 0482), L'Hospitalet de Llobregat, Catalonia
  - Clinica Universidad de Navarra-Hematology Department ( Site 0485), Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal-Hematology ( Site 0484), Madrid, Madrid, Comunidad de
  - Hospital Costa del Sol-Hematology Service ( Site 0493), Marbella, Malaga
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 0489), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 0494), Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca-Hematology ( Site 0488), Salamanca
- Sweden (5):
  - Skånes Universitetssjukhus Lund-Department of Hematology ( Site 0544), Lund, Skåne County
  - Karolinska Universitetssjukhuset Huddinge ( Site 0541), Huddinge, Stockholm County
  - Akademiska sjukhuset ( Site 0545), Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset-Department of hematology and coagulation ( Site 0543), Gothenburg, Västra Götaland County
  - Universitetssjukhuset Örebro ( Site 0542), Örebro, Örebro County
- Taiwan (4):
  - Chang Gung Memorial Hospital- Chiayi ( Site 0242), Chiayi City, Chiayi
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 0245), Tainan
  - National Taiwan University Hospital ( Site 0241), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0243), Taoyuan District
- Turkey (Türkiye) (10):
  - Ege Universitesi Hastanesi ( Site 0503), Bornova, İzmir
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi-Hemotology ( Site 0510), Ankara
  - Hacettepe Universite Hastaneleri-Department of Hematology ( Site 0505), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 0502), Ankara
  - Ankara UTF Cebeci Arastırma ve Uygulama Hastanesi ( Site 0511), Ankara
  - Antalya Egitim ve Arastırma Hastanesi ( Site 0508), Antalya
  - Trakya University Medical Faculty Hospital-Hematology ( Site 0501), Edirne
  - Medipol Mega Universite Hastanesi ( Site 0504), Istanbul
  - Kocaeli Üniversitesi-Hematology ( Site 0506), Kocaeli
  - Ondokuz Mayıs Universitesi-hematology ( Site 0507), Samsun
- United Kingdom (9):
  - Glan Clwyd Hospital ( Site 0528), Bodelwyddan, Denbighshire
  - Gloucestershire Royal Hospital ( Site 0521), Gloucester, Gloucestershire
  - Lincoln County Hospital ( Site 0535), Lincoln, Great Britain
  - Boston Pilgrim Hospital ( Site 0525), Boston, Lincolnshire
  - University College London Hospital ( Site 0527), London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust ( Site 0523), London, London, City of
  - Hammersmith Hospital ( Site 0533), London, London, City of
  - Freeman Hospital ( Site 0532), Newcastle upon Tyne
  - Royal Gwent Hospital ( Site 0524), Newport

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26132&tenant=MT_MSD_9011